CLINICAL TRIAL: NCT00868400
Title: Multi-centre Double-blind Randomized Trial of the Clinical Value of Preoperative Oral Carbohydrate Loading in Colorectal Surgery.
Brief Title: Clinical Value of Preoperative Oral Carbohydrate Loading in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Collaborators: General Hospital of Nikaia "Saint Panteleimon" (Other); University Clinical Centre of Kosova (Other); University Hospital, Ghent (Other); Szeged University (Other); European Society for Surgical Research (Other)
Responsible Party: Principal Investigator, Mehmet Fatih Can, Associate Professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRECALICS
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Disorders; Colorectal Surgery
Keywords: Preoperative care; colorectal surgery; carbohydrate; fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): High-carbohydrate
  Interventions: Dietary Supplement: commercially available high-carbohydrate beverage
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: flavored water
- 3 (No Intervention): Control

INTERVENTIONS:
Dietary Supplement: commercially available high-carbohydrate beverage — 800 ml before the day of surgery, and additional 400 ml two hours prior to surgery
  Arms: 1
Dietary Supplement: flavored water — will be given in doses equal to those of high-carbohydrate beverage
  Arms: 2

SUMMARY:
The aim of this study is to provide conclusive clinical evidence as to whether or not the preoperative administration of oral carbohydrate-rich solutions is effective on the outcomes of patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
Preoperative oral carbohydrate loading is an issue that has been investigated extensively in terms of its fundamental and biochemically apparent effects and potential benefits. Most commonly, proponents of the application advocate that it may be beneficial for improving patient outcomes and for decreasing complication rate by attenuating postoperative insulin resistance. To date, however, no study with a sufficient sample size has been able to demonstrate that it has a marked value in clinical practice. Almost all of the clinical benefits ascribed to the application have been based on subjective well-being, which can also be provided with non specific simple beverages. A study conducted to show whether or not the application has direct influence on patient outcome, therefore, could significantly contribute insights on this topic. The present study was planned to consist of three study arms, namely: 1.Study group, which will be given high-carbohydrate beverage (Nutricia preOp®, Numico, Zoetermeer, The Netherlands) 2. Placebo group, which will be given flavored water, and 3. Control group (surgery after overnight fast). The revised power analysis shows that an accrual of 74 patients in each group would allow detecting a 15% difference in the rate of complications with 80% power at the 5% level of significance (two tailed). We hope we will have recruited at least 220 subjects at the end of a two-year course. Once the data recording is complete, this study will be the largest one ever conducted to investigate this topic.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing colorectal surgery for malignant or benign diseases

Exclusion Criteria:

* diabetes
* disorders that prolongs gastric emptying
* existence of an increased risk for aspiration of gastric content
* anal surgery (haemorrhoidectomy, fistulotomy...etc)
* emergency operations

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Overall 30-day complication rate | 2 years

SECONDARY OUTCOMES:
Patient discomfort | 2 years
need for insulin infusion | 2 years
Length of intensive care unit and hospital stay | 2 years
Patient recovery | 2 years
Overall 30-day mortality rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet F Can, Assist Prof, Study Director — Gulhane School of Medicine, Department of Surgery; Avdyl Krasniqi, MD, PhD, Principal Investigator — University Clinical Centre of Kosova, Department of Surgery; Costas Vagianos, Assoc Prof, Principal Investigator — Agios Panteleimon Regional Hospital, Deparment of Surgery; Gokhan Yagci, Assoc Prof, Principal Investigator — Gulhane School of Medicine, Department of Surgery; Gyorgy Lazar, Prof, Principal Investigator — University of Szeged, Department of Surgery; Wim P Ceelen, MD, PhD, Prof, Principal Investigator — Ghent University Hospital, Department of Surgery
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)